CLINICAL TRIAL: NCT04025853
Title: Inflammatory Biomarkers to Diagnose and Monitor Diabetic Foot Osteomyelitis
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Larry Lavery, Professor, Plastic Surgery; Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: 042015-048
Record Dates: First submitted 2019-05-17; First posted 2019-07-19 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to do a retrospective chart review of 500 patients admitted to the hospital between January 1, 2010 and December 31, 2015 with diabetic foot infections. The investigators will define a positive case of osteomyelitis as bone with positive bacterial cultures or histologic finding of acute or chronic osteomyelitis. Levels of inflammatory biomarkers (CRP, ESR) will be collected from the charts from the first time of diagnosis. Because wound healing, biomarker levels and resolution of infection are clearly affected by other factors such as demographics, medical/surgical history, social history, medications, laboratory results, peripheral arterial disease, wound severity, and treatment factors such as type of antibiotics, off-loading, debridement and vascular surgery interventions these will also be collected. The investigators will collect this clinical data for both cohorts.

DETAILED DESCRIPTION:
Introduction and Purpose:

Foot infections are one of the most common reasons for hospitalization and amputation in persons with diabetes. It is often difficult to determine if diabetic foot ulcers have osteomyelitis. Inaccurate diagnosis of osteomyelitis leads to unnecessary antibiotic treatment, surgery, and amputation. In addition, there are no good diagnostic tests to determine when osteomyelitis has been successfully treated. The results of medical treatment for DFO alone are poor with success rates of 60%.

The investigators plan a retrospective chart review of 500 patients admitted to our hospital between January 1, 2010 and December 31, 2015 with diabetic foot infections. We will define diabetic foot osteomyelitis as bone with positive bacterial cultures or histologic finding of acute or chronic osteomyelitis.

The investigators also plan to review 200 foot infections in non-diabetics.

Specific Aims Aim 1. Evaluate the effectiveness of biomarkers to diagnose diabetic foot osteomyelitis using bone culture and histopathology as the "gold standard" to establish the diagnosis.

Aim 2. Evaluate the effectiveness of biomarkers to differentiate osteomyelitis from deep soft tissue infections in patients with diabetic foot ulcers.

There is no risk to subjects, except a minimal risk of Loss of Confidentiality. Information gained from the analysis of data may lead to a better understanding of the mechanisms of diabetic ulcer formation and DFO and inform future research to develop better treatments.

Background:

There is a worldwide epidemic of diabetes. According to data from the World Health Organization, the world prevalence of diabetes among adults was 6.4% in 2010, affecting 285 million adults worldwide. The prevalence of diabetes is expected to increase to 7.7% by 2030 (439 million adults) [1]. In the United States, the prevalence of diabetes increased by 26% from 2007 to 2012, and the associated cost of managing this disease increased from $174 to $245 billion (41% increases) in the same time period [2]. The U.S. Centers for Disease Control and Prevention estimate that 26 million people in the US have diabetes [3]. By 2034 this is expected to increase to 44 million people [4]. Diabetic foot infections are a common, costly, and life altering complication.

As part of the worldwide epidemic of diabetes mellitus, the prevalence of lower extremity complications is rising. Patients with diabetes are now confronted with a 25% lifetime risk of developing a foot ulcer. Among persons with diabetes, foot infections are one of the most common reasons for hospitalization and lower extremity amputations. 20% of all patients with infected foot ulcers end up with amputation of the foot or leg; however, when there is osteomyelitis, the risk of amputation increases 3 fold. On average patients with diabetic foot osteomyelitis have longer hospitalizations (32 vs.14 days), more surgeries (65% vs. 31%), and longer treatment with intravenous antibiotics (32 vs. 14 days) compared to patients with soft tissue infections.

Diagnosing diabetic foot osteomyelitis (DFO) and monitoring resolution of infection remains a challenge with very little evidence that biomarkers or imaging techniques can accurately assess the presence of bone infection. Bone culture and histology are considered to be the gold standard in most guidelines to diagnose DFO but it is not routinely done in clinical practice. The erythrocyte sedimentation rate (ESR) has been suggested to be the best currently available laboratory test to diagnose and monitor DFO. Only a few small studies have evaluated the value of C-reactive protein (CRP) to diagnose and monitor osteomyelitis in the diabetic foot. Unfortunately, the level of quality of the available studies is low, patient populations are small and the heterogeneous use of reference tests to confirm DFO make it difficult to compare data.

Preliminary Studies:

Preliminary data suggest that CRP is a valuable marker to distinguish bone infection in patients with diabetic foot ulcers. Also, results show that ESR and CRP may be helpful when monitoring success of therapy. The investigators hypothesize that CRP will be the most valuable marker to diagnose diabetic foot osteomyelitis and that ESR gives the clinician more information during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the investigators.
* Male and female
* ages 18-89
* moderate diabetic foot infections (according to IDSA criteria) and non-diabetic foot infections who presented for treatment between January 1, 2010 and December 31, 2015. •positive case of osteomyelitis as bone with positive bacterial cultures or histologic finding of acute or chronic osteomyelitis.
* The investigators will only enroll patients who have an initial baseline CRP or ESR within 72 hours of admission, before any surgical procedures.

Exclusion Criteria:

•Not meeting inclusion criteria.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with foot infections.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of biomarkers to diagnose diabetic foot osteomyelitis using bone culture and histopathology as the "gold standard" to establish the diagnosis. | 2 years
  To correlate the level of white blood cell count, c-reactive protein and erythrocyte sedimentation rate with the results of bone culture and histopathology as the "gold standard" to establish the diagnosis.
Evaluate the effectiveness of biomarkers to differentiate osteomyelitis from deep soft tissue infections in patients with diabetic foot ulcers. | 2 years
  To correlate the accuracy of white blood cell count, c-reactive protein and erythrocyte sedimentation rate to differentiate osteomyelitis by observing the results of bone culture and histopathology as the "gold standard" to establish the diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guariguata L, Whiting D, Weil C, Unwin N. The International Diabetes Federation diabetes atlas methodology for estimating global and national prevalence of diabetes in adults. Diabetes Res Clin Pract. 2011 Dec;94(3):322-32. doi: 10.1016/j.diabres.2011.10.040. Epub 2011 Nov 17. PMID 22100977
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086
- [Background] Huang ES, Basu A, O'Grady M, Capretta JC. Projecting the future diabetes population size and related costs for the U.S. Diabetes Care. 2009 Dec;32(12):2225-9. doi: 10.2337/dc09-0459. PMID 19940225
- [Background] Lipsky BA, Berendt AR, Deery HG, Embil JM, Joseph WS, Karchmer AW, LeFrock JL, Lew DP, Mader JT, Norden C, Tan JS; Infectious Diseases Society of America. Diagnosis and treatment of diabetic foot infections. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):212S-238S. doi: 10.1097/01.prs.0000222737.09322.77. PMID 16799390